CLINICAL TRIAL: NCT05681429
Title: Accelerated Recovery Following Opioid-free Anaesthesia in Supratentorial Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Dr. Chu Mei Yeen, Principal Investigator, Trainee in Master of Anaesthesiology & Intensive Care, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022724-11404
Record Dates: First submitted 2022-12-06; First posted 2023-01-12 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Opioid-Free Anaesthesia
Keywords: Opioid-free Anaesthesia; Supratentorial Craniotomy; Accelerated recovery
MeSH Terms: interventions — Lidocaine; Dexmedetomidine; Sevoflurane; Acetaminophen; parecoxib

STUDY DESIGN:
Intervention Model Description: Single-blinded prospective randomised controlled trial
Who Masked: Participant
Masking Description: Single-blinded RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-based Anaesthesia (Placebo Comparator): This arm will be given drugs for standard opioid-based anaesthesia.
  Interventions: Drug: Lignocaine, Dexmedetomidine, Sevoflurane, Paracetamol, Parecoxib
- Opioid-free Anaesthesia (Experimental): This experimental arm will be given drugs for opioid-free anaesthesia as stated below to replace opioids used:
  Intravenous (IV) Lignocaine (1.5 mg/kg) Intravenous Infusion (IVI) Dexmedetomidine (0.2-0.7 mcg/kg/h) & volatile (sevoflurane) ~ Minimum Alveolar Concentration (MAC) 0.9-1.0 IV Paracetamol 1 gm (give after scalp block) IV Parecoxib 40 mg (give 30 minutes before end of surgery) IV Ondansetron 4 mg (give 30 minutes before end of surgery) IV Metoclopramide 10 mg (rescue)
  Interventions: Drug: Lignocaine, Dexmedetomidine, Sevoflurane, Paracetamol, Parecoxib

INTERVENTIONS:
Drug: Lignocaine, Dexmedetomidine, Sevoflurane, Paracetamol, Parecoxib — To compare the recovery outcome of patients who undergo supratentorial craniotomy with opioid-based anaesthesia and opioid-free anaesthesia
  Other Names: Group B

SUMMARY:
Anaesthesia for craniotomy (open skull/brain) surgery focuses on maintaining blood supply to brain, avoiding factors that may lead to increased pressure in brain and aim for early neurological recovery. In recent decades, opioids have always been a mainstay for pain management and opioid-based anaesthesia (OBA). However, opioid use poses a significant number of adverse effects such as breathing depression, prolonged sedation, nausea and vomiting, itchiness, and many more. In view of this, recent studies on anaesthesia for craniotomy has noted a paradigm shift towards opioid-sparing or opioid-free anaesthesia (OFA) to prevent opioid-related adverse effects which might prolong patients' recovery. In order to guide anaesthesiologists' dosing of hypnotics and analgesics to provide appropriate depth of anaesthesia and adequate pain control, as well as to prevent under or overdosing, CONOX monitor is used during operation to measure depth of anaesthesia and painful stimulus.

This clinical study will take place in neurosurgical operation theatres and neurosurgical intensive care unit (ICU) of University of Malaya Medical Centre (UMMC), Kuala Lumpur, Malaysia.

DETAILED DESCRIPTION:
Anaesthesia for craniotomy surgery focuses on maintaining cerebral perfusion, avoiding factors that may lead to increased intracranial pressure and aim for early postoperative neurological recovery. In recent decades, opioids have always been a mainstay for perioperative pain management and play an important role as the standard of care - opioid-based anaesthesia (OBA). However, opioid use poses a significant number of adverse effects such as respiratory depression, prolonged sedation, postoperative nausea and vomiting (PONV), pruritus, ileus, urinary retention, and hyperalgesia. This should be avoided in patients who undergo craniotomy as they can lead to an inaccurate neurological examination because of excessive sedation and have the potential to mask early signs of intracranial complications. Besides, opioid-induced respiratory depressions cause hypercapnia which increases cerebral blood flow and may lead to cerebral oedema. Opioid-induced PONV leads to a spike in intracranial pressure which can be detrimental for post-craniotomy patients. Despite this, adequate pain management is vital as suboptimal pain control drives sympathetic efflux, promoting hypertension that may increase morbidity and mortality through intracranial haemorrhage. In view of this, recent studies on anaesthesia for craniotomy has noted a paradigm shift towards opioid-sparing or opioid-free anaesthesia (OFA) to prevent opioid-related adverse effects which might prolong patients' recovery post-craniotomy. Multi-modal analgesia is also incorporated in many practices nowadays to achieve optimal intraoperative and post-craniotomy pain control. In order to guide anaesthesiologists' dosing of hypnotics and analgesics to provide appropriate depth of anaesthesia and adequate pain control, as well as to prevent under or overdosing, CONOX monitor might be used intraoperatively to measure hypnotic effect (qCon) and probability of response to noxious stimulus (qNox).

This prospective randomised controlled trial clinical study will take place in neurosurgical operation theatres and neurosurgical intensive care unit (ICU) of University of Malaya Medical Centre (UMMC), Kuala Lumpur, Malaysia to compare intraoperative and postoperative outcomes of patients who undergo elective supratentorial craniotomy with opioid-free anaesthesia (OFA) and those with opioid-based anaesthesia (OBA).

ELIGIBILITY:
Inclusion Criteria

* Adult patients who have supratentorial lesions going for elective craniotomies (age group- 18-65 years old)
* Patients with Glasgow Coma Scale of 15 (E4V5M6)
* Patients who are fit to give consent
* Power of elbow flexion of patient's dominant hand score 5 with Medical Research Council (MRC) Muscle scale
* American Society of Anaesthesiologists (ASA) Physical Status Classification I - III patients

Exclusion Criteria

* Patients who refused or not fit to consent for participation
* Patients with Glasgow Coma Scale less than 15
* Patients who have known allergy to the drugs used in this study
* Patients on chronic opioid use (Chronic opioid use is defined as having any number of opioid prescriptions or dosing for at least 90 days continuously)
* Patients going for emergency craniotomies for supratentorial lesions
* Patients who are not fit for extubation postoperatively
* Patients with chronic kidney disease Stage 3A and above (eGFR less than 60 ml/min/1.73m2)
* Patients with known case of liver cirrhosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
To compare sedation score of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From the time of arrival in peri anaesthesia care unit till 24 hours post time of end of surgery
  Modified Ramsay Sedation Score, minimum score: 1, maximum score: 8, the lower the score, the better the conscious level

SECONDARY OUTCOMES:
To compare time to extubation of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From time of cessation of anaesthetic agents (remifentanil/sevoflurane/dexmedetomidine) till time of removal of endotracheal tube, up till 24 hours
  Time to Extubation in minutes , the shorter the duration of time, the better the recovery outcome
To compare pain score of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From time of arrival in peri anaesthesia care unit till 24 hours post time of end of surgery
  Numerical Pain Score , minimum score: 0, maximum score: 10, the lower the pain score,the better the pain control
To compare time to first rescue of opioid analgesia of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From time of arrival in peri anaesthesia care unit till time to first recuse opioid analgesia is administered, up till 24 hours
  Time to first rescue of opioid analgesia (fentanyl) in minutes
To compare time to Modified Ramsay Sedation Score of 2 of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From time of arrival in peri anaesthesia care unit till Modified Ramsay Sedation Score of 2, up till 24 hours
  Time to Modified Ramsay Sedation Score of 2 in minutes, the shorter the duration of time, the better the recovery outcome
To compare Short Orientation Memory Concentration Test (SOMCT) score of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From time of arrival in peri anaesthesia care unit till completion of Short Orientation Memory Concentration Test (SOMCT), up till 24 hours
  Short Orientation Memory Concentration Test (SOMCT) score, minimum score: 0, maximum score: 28, the higher the score, the better the cognitive function
To compare time to return of power of elbow flexion of dominant hand to 5 of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From time of arrival in peri anaesthesia care unit till time to return of power of elbow flexion of dominant hand to 5, up till 24 hours
  Time to return of Power of elbow flexion of dominant hand to 5 in minutes, the shorter the duration of time, the better the recovery of muscle power
To compare modified Aldrete score of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From time of arrival in peri anaesthesia care unit till discharge from peri anaesthesia recovery unit, up till 24 hours
  Modified Aldrete score, minimum score: 0, maximum score: 10, the higher the score, the better the recovery
To compare duration of stay in peri anaesthesia care unit (PACU) of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From the time of arrival in peri anaesthesia care unit till discharge from peri anaesthesia recovery unit, up till 24 hours
  Duration of stay in peri anaesthesia care unit (PACU) in minutes, the shorter the duration of stay, the better the recovery outcome
To compare total postoperative opioid consumption of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From the time of arrival in peri anaesthesia care unit till 24 hours post time of end of surgery
  Total postoperative opioid consumption (in morphine equivalent- in milligram), the lower the opioid consumption, the better the pain control
To compare incidence of postoperative nausea and vomiting (PONV) of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From the time of arrival in peri anaesthesia care unit till 24 hours post time of end of surgery
  Incidence of postoperative nausea and vomiting (PONV), yes or no
To compare total length of hospital stay of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From the day of admission to hospital till the day of discharge from hospital, up till 365 days
  Length of hospital stay in days, the shorter the number of days of hospital stay, the better the recovery outcome
To compare haemodynamic responses: Blood Pressure during intubation of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of induction of anaesthesia till end of intubation process
  Haemodynamics readings: Blood Pressure (mmHg)
To compare haemodynamic responses: Heart Rate during intubation of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of induction of anaesthesia till end of intubation process
  Haemodynamics readings: Heart Rate (beats per minute)
To compare haemodynamic responses: Mean Arterial Pressure during intubation of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of induction of anaesthesia till end of intubation process
  Haemodynamics readings: Mean Arterial Pressure (MAP) (mmHg)
To compare haemodynamic responses : Blood Pressure during cranial pinning of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of cranial pinning till end of cranial pinning process
  Haemodynamics readings: Blood Pressure (mmHg)
To compare haemodynamic responses: Heart Rate during cranial pinning of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of cranial pinning till end of cranial pinning process
  Haemodynamics readings: Heart Rate (beats per minute)
To compare haemodynamic responses: Mean Arterial Pressure during cranial pinning of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of cranial pinning till end of cranial pinning process
  Haemodynamics readings: Mean Arterial Pressure (MAP) (mmHg)
To compare haemodynamic responses: Blood Pressure during skin incision of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of skin incision till end of skin incision process
  Haemodynamics readings: Blood Pressure (mmHg)
To compare haemodynamic responses : Heart Rate during skin incision of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of skin incision till end of skin incision process
  Haemodynamics readings: Heart Rate (beats per minute)
To compare haemodynamic responses: Mean Arterial Pressure during skin incision of patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of skin incision till end of skin incision process
  Haemodynamics readings: Mean Arterial Pressure (MAP) (mmHg)
To compare the difference of qCon and qNox indexes using CONOX in patients who undergo elective supratentorial craniotomies with opioid-free anaesthesia and those with opioid-based anaesthesia. | From start of induction of anaesthesia till end of surgery
  qCON and qNOX readings from CONOX monitor, minimum value: 0, maximum value: 100, optimum value intraoperatively: 40-60, the higher the score, the more higher the level of alertness of patient

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jeyaganesh a/l S. Veerakumaran, Study Chair — University of Malaya
Locations (1):
- Universiti Malays Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Research data WITHOUT participants' personal information and identifier will be shared with other researchers
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Dec 2023 till Dec 2024
Access Criteria: Research data WITHOUT participants' personal information and identifier will be shared with other researchers

DOCUMENTS (1):
  • Informed Consent Form (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT05681429/ICF_000.pdf